CLINICAL TRIAL: NCT06783738
Title: Assessing Fitness, Physical Activity and Leukocyte Genomic Response to Exercise in Acute Lymphoblastic Leukemia (ALL) Patients in Remission
Brief Title: Physical Activity in Acute Lymphoblastic Leukemia (ALL)
Acronym: ALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Shlomit Aizik, Professor, University of California, Irvine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1519
Record Dates: First submitted 2024-05-03; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Acute Leukemia
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy (Active Comparator): Aerobic fitness will be assessed using incremental cycle-ergometer exercise test to determine peak maximum rate of oxygen use (VO2) in healthy subjects. Exercise testing will be performed at the University of California Irvine (UCI) Pediatric Exercise and Genomics Research Center (PERC)/Institute for Clinical and Translational Science (ICTS) Applied Physiology/Human Performance Core Laboratory. The work rate will increase by 5-10 W per min (or adjusted according to the subject's age and fitness level) so that the total exercise time will roughly equal 8-12 min, and each subject will exercise to the limit of his or her tolerance.
  Interventions: Other: Exercise
- Children Diagnosed with ALL (Experimental): Aerobic fitness will be assessed using incremental cycle-ergometer exercise test to determine peak maximum rate of oxygen use (VO2) in ALL patients. Exercise testing will be performed at the University of California Irvine (UCI) Pediatric Exercise and Genomics Research Center (PERC)/Institute for Clinical and Translational Science (ICTS) Applied Physiology/Human Performance Core Laboratory. The work rate will increase by 5-10 W per min (or adjusted according to the subject's age and fitness level) so that the total exercise time will roughly equal 8-12 min, and each subject will exercise to the limit of his or her tolerance.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The participants will come to our lab twice. In the first visit we will perform a fitness assessment, using a noninvasive, cardiopulmonary exercise testing used routinely to measure fitness in children.

SUMMARY:
Acute lymphoblastic leukemia (ALL) is the most common blood cancer of children and adolescents. Remarkable progress has been made in treating this deadly disease, but many children suffer relapses despite these advances. There are mounting data showing that lifestyle factors, specifically levels of exercise and nutritional intake, can have measurable and substantial impact on how well patients with a variety of cancers respond to treatment. It is not surprising that children and adolescents who have survived ALL tend to exercise less and be less fit than otherwise healthy subjects. But very little is known in pediatric patients with ALL about how exercise might be beneficial and prolong disease-free intervals. Recently, the National Cancer Institute (NCI) put out a call for research proposals designed to test mechanisms through which lifestyle interventions like exercise might prolong survivorship in cancer patients. The NCI specifically stressed the need to better understand the biological mechanisms through which behaviors like exercise could benefit cancer patients.

Exciting work in our laboratory (HS# 2002-2598) demonstrates the substantial effect that exercise has on white blood cell gene expression. Our data actually suggest heretofore undiscovered mechanisms that might explain why exercise might be beneficial for children and teenagers treated with ALL.

Under under HS#2012-9248, 8 pediatric ALL patients and 7 healthy controls, will be tested (for an overall sample size of 15) with, cardiopulmonary exercise testing used routinely to measure fitness in children. These data will provide us with essential information about fitness, and the immune system response to exercise in these patients and will be used to develop a broader set of studies and exercise interventions that, hopefully, will identify the ways in which exercise can serve as an adjunct to standard therapy for children with ALL.

DETAILED DESCRIPTION:
Acute lymphocytic leukemia (ALL) is the most common hematological malignancy in children and adolescents. The gratifying and dramatic improvement in the survivorship of ALL is a testament to the strength of collaborative, multidisciplinary translational research efforts. Yet many gaps in our fundamental knowledge of disease mechanisms in ALL remain and hamper our ability to prolong remission and decrease disease relapse. There is increasing evidence that environmental, lifestyle factors such as physical exercise and fitness may play a beneficial role in cancer survivorship. The NCI has recently posted a Program Announcement to stimulate research on the impact of lifestyle interventions (e.g., exercise, nutrition) on cancer survivorship. The goal of this project is a development of a series of novel, hypothesis-driven proof of concept studies to explore ways in which exercise might benefit survivorship in ALL. The purpose of this initial project and Institutional Review Board (IRB) application is to gather minimally invasive data about patterns of physical activity and exercise, and leukocyte genomic response to exercise in children treated for ALL. These data will be essential in developing a larger protocol in response to the National Cancer Institute Program Announcement (NCI PA), one that addresses the NCI challenge that, "The biobehavioral mechanisms and pathways through which lifestyle interventions may increase survival following cancer are unknown." In addition, a number of studies have demonstrated that cardiovascular risk factors (such as BMI) in ALL survivors deteriorate following therapy. Exercise training interventions can improve cardiovascular risk in these patients; however, are difficult to implement in this population.

Consequently, in preparation for a larger study of exercise training on leukocyte genomic and epigenetic responses in ALL survivors, an essential biobehavioral component of any training study will be tested, namely, readiness for exercise training using approaches developed by researchers in our group. This part of our research will help us identify and target the unique set of fears and obstacles that almost invariably accompany children and adolescents (and their caregivers) who survive life-threatening diseases.

ELIGIBILITY:
Inclusion Criteria:

* Ages 10-17 (males and females)
* Diagnosed with ALL in remission stage
* No evidence of disability that would impair participation in a vigorous physical activity challenge

Exclusion Criteria:

* Pregnancy or breastfeeding
* Use of illegal drugs or alcohol
* Other conditions that preclude exercise (such as neuromotor disease, heart disease, or any other condition that would prevent a child from participating in vigorous physical activity)

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2003-01-31 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Gene Expression Profile (RNAseq) | 8-12 minutes
  Gene expression profile before and after acute exercise in children with acute lymphoblastic leukemia in remission compared to healthy control. Differential gene expression analysis was performed using DESeq2 (v.1.38.3). Paired design was used to account for samples from the same patient. Multifactor design with interaction terms was applied for group differences.

SECONDARY OUTCOMES:
Natural Killer (NK) Activity (NKCA) | Baseline and immediately following acute exercise
  NKCA before and after acute bout of exercise in ALL children and healthy controls. NKTEST® kit from Glycotope Biotechnology (Allele Biotechnology, San Diego, CA) was used to evaluate NKCA per the kit instructions. The NKTEST kit quantifies NKCA using green fluorescent. NKCA was reported as the percentage of red-stained cells over total green-stained cells.

CONTACTS AND LOCATIONS:
Overall Officials: Shlomit Radom-Aizik, Ph.D., Principal Investigator — University of California, Irvine Pediatric Exercise and Genomics Research Center (PERC)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esbenshade AJ, Simmons JH, Koyama T, Koehler E, Whitlock JA, Friedman DL. Body mass index and blood pressure changes over the course of treatment of pediatric acute lymphoblastic leukemia. Pediatr Blood Cancer. 2011 Mar;56(3):372-8. doi: 10.1002/pbc.22782. PMID 20860019
- [Background] Jarvela LS, Niinikoski H, Lahteenmaki PM, Heinonen OJ, Kapanen J, Arola M, Kemppainen J. Physical activity and fitness in adolescent and young adult long-term survivors of childhood acute lymphoblastic leukaemia. J Cancer Surviv. 2010 Dec;4(4):339-45. doi: 10.1007/s11764-010-0131-0. Epub 2010 Jun 15. PMID 20552291
- [Background] Hartman A, Hop W, Takken T, Pieters R, van den Heuvel-Eibrink M. Motor performance and functional exercise capacity in survivors of pediatric acute lymphoblastic leukemia. Pediatr Blood Cancer. 2013 Mar;60(3):494-9. doi: 10.1002/pbc.24243. Epub 2012 Jun 28. PMID 22745035
- [Background] Jarvela LS, Kemppainen J, Niinikoski H, Hannukainen JC, Lahteenmaki PM, Kapanen J, Arola M, Heinonen OJ. Effects of a home-based exercise program on metabolic risk factors and fitness in long-term survivors of childhood acute lymphoblastic leukemia. Pediatr Blood Cancer. 2012 Jul 15;59(1):155-60. doi: 10.1002/pbc.24049. Epub 2011 Dec 19. PMID 22184098
- [Background] Hartman A, te Winkel ML, van Beek RD, de Muinck Keizer-Schrama SM, Kemper HC, Hop WC, van den Heuvel-Eibrink MM, Pieters R. A randomized trial investigating an exercise program to prevent reduction of bone mineral density and impairment of motor performance during treatment for childhood acute lymphoblastic leukemia. Pediatr Blood Cancer. 2009 Jul;53(1):64-71. doi: 10.1002/pbc.21942. PMID 19283791